CLINICAL TRIAL: NCT02566681
Title: Phase I Clinical Trial of Use of Autologous Bone Marrow Stem Cells Seeded on Porous Tricalcium Phosphate Matrix and Demineralized Bone Matrix in Patients With Osteonecrosis (MSC/ONM)
Brief Title: Clinical Trial of Use of Autologous Bone Marrow Stem Cells Seeded on Porous Tricalcium Phosphate Matrix and Demineralized Bone Matrix in Patients With Osteonecrosis
Acronym: MSC/ONM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Instituto Murciano de Investigación Biosanitaria Virgen de la Arrixaca (Other); Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other); Hospital Universitario Virgen de la Arrixaca (Other); Spanish National Health System (Other); Public Health Service, Murcia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC/ONM; 2012-005813-38 (EudraCT Number)
Record Dates: First submitted 2015-01-30; First posted 2015-10-02 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Osteonecrosis of Jaw

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSC construct for Osteonecrosis (Experimental): Patients with definite diagnosis of osteonecrosis of the jaw by clinical and radiological examination of any etiology will receive a construct made of Bone Marrow Stem Cell + Tricalcium Phosphate + Demineralized Bone Matrix (MSC+TP+DBM).
  Interventions: Biological: MSC construct for Osteonecrosis

INTERVENTIONS:
Biological: MSC construct for Osteonecrosis — 30 days before implanting the construct made with MSC + TP + DBM, bone marrow of patients diagnosed with osteonecrosis of the jaw included in the clinical trial is obtained. The bone marrow will be obtained according to standard practice for Hematologists of the Haematology University Hospital Virgen de la Arrixaca (HCUVA).
  Mononuclear bone marrow cells were separated and cultured in GMP conditions (Good Manufacturing Practices). The cells are seeded on tricalcium phosphate and maintained in culture for 14 days.
  The day when the implant is performed, the patient is prepared in the operating room. The area where the implant will be placed is cleaned. Mesenchymal cells seeded in tricalcium phosphate are mixed with demineralized bone matrix and It's coagulated with autologous platelet rich plasma and grafting is performed. Finally, the oral mucosa or skin will be sealingly closed by silk sutures.

SUMMARY:
The purpose of this study is to evaluate the safety of use of autologous bone marrow stem cells seeded on porous tricalcium phosphate matrix and demineralized bone matrix in patients with osteonecrosis of the jaw by a prospective, single-center, open, nonrandomized and unblinded clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mandibular osteonecrosis of any etiology defined by clinical and radiological examination.
* Bone defect anteroposterior dimension less than or equal to 4 cm in the mandible or the maxilla 2.5, and / or bone bed sufficient to ensure the integrity of the construct during surgery.
* No response to conservative treatment.
* Provide sufficient assurance of adherence to protocol.
* Provide written consent
* Meet all the inclusion criteria

Exclusion Criteria:

* Concomitant psychiatric illness.
* Uncontrolled concomitant systemic disease.
* Active infectious disease in the focus of mandibular osteonecrosis.
* Neoplastic disease in complete remission less than 2 years.
* Pregnant patients.
* Patients with active feeding.
* Patients physically fertile, defined as all women physiologically capable of becoming pregnant, UNLESS they are using reliable methods of contraception.
* Patients with cardiac disease, renal, hepatic, systemic, immune that may influence patient survival during the test.
* Inclusion in other clinical trials in active treatment.
* Inability to understand the informed consent.
* You need not meet any exclusion criteria

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Rate of serious adverse events related to the procedure. | 24 months from baseline
  Apparition of Bone ischemic events. Neoformations.
Rate of non-serious adverse events related to the procedure. | 24 months from baseline
  Local infection of the surgical wound. Pseudarthrosis implant. Allergic reactions.

SECONDARY OUTCOMES:
Time to Repair the injury | 24 months from baseline
Local pain assessed by visual analog scale | 24 months from baseline
Bone formation, measured by Computed tomography (mm) | 24 months from baseline
Quality of life, measured by EuroQol-5D. | 24 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Victor Villanueva San Vicente, MD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca; Francisco J Rodríguez Lozano, PhD, Principal Investigator — Universidad de Murcia
Locations (1):
- Hospital Clínico Virgen de la Arrixaca, El Palmar, Murcia, Spain